CLINICAL TRIAL: NCT05980754
Title: Clinical Study on Exploring High Risk Factors Inducing the Progress of Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dongyang Liu, Principal Investigator, Peking University Third Hospital
Other Study IDs: DCTC-IIR202305
Record Dates: First submitted 2023-04-17; First posted 2023-08-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: T2D

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy group: No intervention
- pre diabetic patients: No intervention
- T2DM patients: No intervention

SUMMARY:
Explore the high related factors of impaired glucose tolerance through descriptive statistics and analysis of variance.

DETAILED DESCRIPTION:
This study is a cross-sectional study planned to include healthy individuals with a BMI within the normal range (18.5<BMI<24 kg/m2) (HbA1c ≤ 5.6%, n=18), pre diabetic patients (5.7% ≤ HbA1c ≤ 6.4%, n=36), and T2DM patients (HbA1c ≥ 6.5%, n=36) among individuals who meet the inclusion criteria and undergo annual physical examinations at the Physical Examination Center of the Third Hospital of Beijing Medical University. Collect the examination values related to demography and glucose metabolism balance of physical examination items, and carry out magnetic resonance imaging (MRI) imaging examination and oral glucose tolerance test (OGTT) results. Explore the high related factors of impaired glucose tolerance through descriptive statistics and analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

• The diagnostic criteria of the American diabetes Association (ADA) were used to determine the type of subjects: Group Healthy individuals: Glycated hemoglobin (HbA1c) ≤ 5.6%; Group Pre T2DM patients: 5.7% ≤ HbA1c ≤ 6.4%; Group T2DM patients: HbA1c ≥ 6.5% (for T2DM patients: this study needs to include first-time or previously diagnosed patients who have not used hypoglycemic drugs within 4 years and HBA1C ≤ 9.5%)Clinical diagnosis of Alzheimer's Disease.

* Male weight ≥ 50kg, female weight ≥ 45kg, 18.5 < BMI < 24kg/m2
* Age range from 40 years old (inclusive) to 65 years old (inclusive), with no less than one-third of either gender
* Subjects voluntarily sign informed consent forms, can maintain good communication with researchers, and comply with the requirements of clinical trials

Exclusion Criteria:

* In the past month and currently taking glucocorticoids, steroids, thiazide diuretics, or atypical antipsychotic drugs
* Some diseases that affect glucose tolerance: type 1 diabetes (T1DM), pancreatic exocrine disease, polycystic ovary syndrome and other endocrine diseases, autoimmune diseases, infection and trauma and other irritability factors
* Diseases that may affect eating: mental illness, post gastrectomy, inflammatory bowel disease, uncontrolled thyroid disease.
* Healthy subjects with a history of gestational diabetes or subjects with direct family members with a family history of diabetes
* Pregnant or lactating women
* Participate in any other clinical trials within 3 months prior to the trial
* Blood donation or loss of ≥ 400mL within 8 weeks before the first cycle of the experiment
* Clinically significant history of ECG abnormalities or family history of long QT syndrome (grandparents, parents, siblings) Suffering from any condition that significantly affects glucose absorption, distribution, metabolism, and excretion within 2 weeks prior to the experiment, or any condition that may pose a hazard to the subject, the detailed conditions are as follows:

  1. History of inflammatory bowel disease, gastritis, ulcers, gastrointestinal or rectal bleeding
  2. A significant history of gastrointestinal surgery (such as gastrectomy, gastroenterostomy, or intestinal resection),
  3. history of pancreatic injury or pancreatitis or clinical evidence, or researchers' judgment of abnormal lipase and amylase,
  4. abnormal liver function tests (such as ALT, AST, serum bilirubin), which are clinically significant, indicate liver disease, cirrhosis, or liver injury. (alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase [ALP], glutamine transpeptidase [GGT], total bilirubin) greater than three times their respective upper limit of normal (ULN).
  5. There is a history or evidence of renal dysfunction, manifested as clinically significant creatinine or urinary composition abnormalities (such as tubular type), or eGFR<60 ml/min/1.73m2
  6. Urinary tract obstruction or difficulty in emptying urine during screening period
* Individuals with any form of medical/implant intolerance, including pacemakers, metal plates, or magnetic resonance imaging (MRI)
* Individuals who have tested positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or syphilis (results within six months are exempt from testing)
* Smokers who smoke more than 10 cigarettes or an equivalent amount of tobacco per day cannot stop smoking during the trial period
* There is a history of drug or alcohol abuse within the 12 months prior to the trial, or evidence of abuse is found during laboratory testing during screening evaluation
* During screening, lying blood pressure (after resting for 5 minutes) exceeds the range of 90-140mm Hg (including 90140) in systolic blood pressure, 50-90 mmHg (including 50, 90) in diastolic blood pressure, or heart rate (HR) exceeds the range of 50 bpm to 100 bpm (including 50100) in heart rate (HR)
* Tumor patients
* Participants are not suitable for the experiment

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Annual physical examination population conducted by the Physical Examination Center of the Third Hospital of Beijing Medical University
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
biochemical parameters including level of Glucose | through study completion, an average of 1 year
  level of Glucose
biochemical parameters including level of C-peptide | through study completion, an average of 1 year
  level of C-peptide
biochemical parameters including level of insulin | through study completion, an average of 1 year
  level of insulin

SECONDARY OUTCOMES:
Liver fat content | 1 year
  magnetic resonance imaging proton density fat fraction (MRI-PDFF)
pancreatic fat content | 1 year
  magnetic resonance imaging proton density fat fraction (MRI-PDFF)

IPD SHARING:
Plan to Share IPD: Undecided